CLINICAL TRIAL: NCT02947503
Title: Pregnancy Outcomes: Effects of Metformin Study (POEM Study), a Long Term Randomized Controlled Study in Gestational Diabetes
Brief Title: Pregnancy Outcomes: Effects of Metformin Study (POEM Study)
Acronym: POEM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bethesda Diabetes Research Center (Other)
Collaborators: Maastricht University Medical Center (Other); University Medical Center Groningen (Other); Frisius Medisch Centrum (Other); Martini Hospital Groningen (Other); Treant Zorggroep (Unknown); Nij Smellinghe Hosptial (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL 2016 POEMS
Record Dates: First submitted 2016-10-20; First posted 2016-10-28 (Estimated); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Gestational Diabetes; Insulin Resistance
Keywords: Gestational Diabetes; Insulin Resistance; Metformin; Hyperinsulinaemia; Prevention of Complications; Long Term Study; Mother and Child; Health Benefits
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance; Hyperinsulinism | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin on top of usual care (Active Comparator): Metformin TEVA 850 mg (1-3 times daily) added to usual care from start of the diagnosis GDM.
  Usual care has been defined as intensive counselling for diet and lifestyle plus insulin therapy if needed.
  Intervention: metformin TEVA 850 mg (1-3 times daily) on top of usual care.
  Interventions: Drug: Metformin TEVA 850 mg
- Usual care (No Intervention): Usual care from start of the diagnosis GDM. Control group without metformin. Usual care has been defined as intensive counselling for diet and lifestyle plus insulin therapy if needed.
  Intervention: usual care.

INTERVENTIONS:
Drug: Metformin TEVA 850 mg — At inclusion, patients (N=500) will be randomized 1:1 to metformin vs usual care (850 mg tablets, 3 times daily or, if tolerance is suboptimal, a lower maximally tolerated dose, 1-2 times daily), on top of diet and lifestyle, with an insulin rescue in both arms if needed.
  Other Names: Metformin
  Arms: Metformin on top of usual care

SUMMARY:
One approach to prevent the rising burden of diabetes is to address the issue of gestational diabetes mellitus (GDM). GDM has a growing prevalence up to 5-10% (and even higher in specific subgroups), with a pregnant population becoming older and more obese worldwide. GDM increases the risks of complications during pregnancy, at delivery and on the longer term, like type 2 diabetes (T2D) and persistent obesity, in mother and child. Moreover, insulin added to diet as the standard care for GDM has disadvantages for mother (maintenance of hyperinsulinaemia, increasing weight and blood pressure) and child (macrosomia, hypoglycaemia) with related adverse pregnancy outcomes. Metformin, as an insulin sensitizer targeting the cause of GDM, may have essential benefits, as suggested by observational studies. However, RCTs with metformin (early positioned in the treatment of GDM) are still lacking. The POEM study is the first Randomized controlled trial (RCT) in GDM to test the hypothesis that metformin, early given from the start of the diagnosis GDM, on top of diet and lifestyle improves clinically relevant pregnancy outcomes in mother and child during pregnancy, at delivery and on the longer term - up to 20 years after birth.

DETAILED DESCRIPTION:
The POEM study was designed to investigate the effects of metformin on top of diet and lifestyle (with insulin rescue if needed) in GDM on eight clinically relevant pregnancy outcomes at delivery, summarized by means of an integrated, newly developed score, the GDM Outcome Score (GOS), and on other relevant outcomes on the longer term in mother and child. The investigators hypothesize that metformin given to women with GDM from the start of the diagnosis reduces risks resulting in relevant health benefits for mother and child during pregnancy, at delivery, and many years thereafter.

The POEM study is a randomized controlled intervention study, consisting of three phases:

* Phase A - from inclusion until six weeks after delivery; intervention study with and without exposure of metformin in mother and (unborn) child: two arms after randomization with 1:1 allocation to Diet + Lifestyle + Metformin (DLM) or Diet + Lifestyle (DL);
* Phase B - from six weeks until 1 year after delivery; intervention study with exposure of DLM vs DL in mother;
* Phase C - from 1 until 20 years after delivery; observational extension study of mother and child without study medication.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with GDM defined as a Fasting Plasma Glucose (FPG) > 5,3 mMol and/or an Oral Glucose Tolerance test (OGTT) with a Plasma glucose (PG) > 7,8 mMol, two hours after the oral intake of 75 gram glucose
* Written informed consent
* Age 18-45 years
* Gestational age at inclusion 16-32 weeks
* Glycohemoglobin test (HbA1c) at inclusion ≤ 48 mmol/mol (6.5% Hb)

Exclusion Criteria:

* Diabetes mellitus before pregnancy, except previous GDM
* Proteinuria: Urine Albumin-to-Creatinine Ratio (UACR) > 35 mg/mmol at screening
* Malignancy during the last 5 years before inclusion, except non-melanoma skin cancer
* Psychiatric and/or mood disorder potentially affecting compliance of treatment
* Chronic liver disease and/or Alanine aminotransferase aspartate transaminase (ASAT) and/or Alanine aminotransferase (ALAT) > 3x Upper Limit of Normal (ULN).
* Chronic renal failure with a Glomerular filtration rate (GFR) < 45 ml/min/1.73m2
* Chronic pulmonary failure with hypoxia
* Significantly uncontrolled hypertension - Systolic blood pressure (SBP) > 160 mm Hg despite medical treatment
* Chronic treatment with corticosteroids
* Intolerance for metformin and/or earlier use of metformin in this pregnancy
* Membership of the POEM study group
* Severe foetal anomaly at inclusion - like major neural tube and/or cardiac malformation
* Ruptured membranes
* Multiple pregnancy
* Inability to understand or read the Dutch language
* Bariatric surgery in medical history
* Hyperemesis gravidarum

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-11-26 (Actual); Primary Completion 2043-12 (Estimated); Study Completion 2043-12 (Estimated)

PRIMARY OUTCOMES:
GDM Outcome Score (GOS) in Phase A | 30 months
  An aggregate score of eight clinically relevant endpoints, as previously defined:
  1. pregnancy related hypertension, including (pre-) eclampsia, according validated guidelines,
  2. large for gestational age baby (LGA) at delivery according validated guidelines,
  3. premature delivery with a gestational age < 37 weeks,
  4. instrumental delivery,
  5. caesarean delivery,
  6. birth trauma, like fractures of clavicle and humerus, subdural / intracerebral haemorrhage,
  7. neonatal hypoglycaemia, defined as blood glucose < 2.6 mmol/l,
  8. admission for neonatal intensive care.
T2D and obesity at the end of Phase B | 42 months
  Incidence of maternal T2DM Weight (kg) and BMI (category) development mother Weight (kg) and BMI (percentile) development child
Development of T2D and obesity during Phase C | 282 months
  Incidence of maternal T2DM Weight (kg) and BMI (category) development mother Weight (kg) and BMI (percentile) development child

SECONDARY OUTCOMES:
Secondary Outcome measures phase A mother | 30 months
  Maternal outcome score (MOS)
  1. Caesarean delivery (yes=1, no=0)
  2. (Pre-)eclampsia, HELPP and PIH (if at least one is diagnosed=yes=1,no=0)
  3. Maternal mortality (yes=1, no=0)
  4. Postpartum haemorrhage (blood loss > 1000 ml)(yes=1, no=0)
  5. Thrombosis (yes=1, no=0)
  For each individual component applies: if occured=1 point. If not occured =0 points. A total score per individual will be calculated (0-5 for MOS). Each component on its own is also a secondary outcome measure.
Secondary Outcome measures phase A child | 30 months
  Neonatal outcome score (NOS)**
  1. IRDS requiring oxygen therapy (CPAP, optiflow, mechanical ventilation or surfactant) (yes=1, no=0)
  2. Stillbirth or neonatal death (yes=1, no=0)
  3. Preterm birth <37 weeks (yes=1, no=0)
  4. Shoulder dystocia (yes=1, no=0)
  5. Instrumental delivery (yes=1, no=0)
  6. Caesarean delivery (yes=1, no=0)
  7. Neonatal hypoglycaemia < 2.6 mml/l (yes=1, no=0)
  8. Neonatal jaundice needing phototherapy (yes=1, no=0)
  9. NICU admission (yes=1, no=0)
  10. Apgar score < 7 at 5 minutes (yes=1, no=0)
  11. Congenital anomaly (to a list, if one anomaly = yes = 1, no=0)
  For each individual component applies: if occured=1. If not occured=0. A total score per individual will be calculated (0-11 for NOS). Each component on its own is also a secondary outcome measure.
  Apgar score as a variable (1-10) at 1, 5, 10 min Foetal weight at delivery in grams
Secondary outcome measures phase B | 42 months
  Hypertension development (yes/no) Thrombotic and CVD events (yes/no) Development of chronic disease (according to list - yes/no)
  Gonadal and gender development (to be determined: question(naires) + potentially additional measurements from research blood panel) Puberty and maturation (to be determined: question(naires) + potentially additional measurements from research blood panel) Educational and intellectual development (levels of education completed) Development of chronic disease (according to list - yes/no)
Secondary outcome measures phase C | 282 months
  Hypertension development (yes/no) Thrombotic and CVD events (yes/no) Development of chronic disease (according to list - yes/no)
  Gonadal and gender development (to be determined: question(naires) + potentially additional measurements from research blood panel) Puberty and maturation (to be determined: question(naires) + potentially additional measurements from research blood panel) Educational and intellectual development (levels of education completed) Development of chronic disease (according to list - yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Adriaan Kooy, Dr., Principal Investigator — BDRC
Locations (4):
- Netherlands (4):
  - Martini hospital Groningen, Groningen
  - University Medical Center Groningen, Groningen
  - Treant Zorggroep, Hoogenveen, Emmen, Stadskanaal
  - Medical Center Leeuwarden, Leeuwarden

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available upon reasonable request. The study protocol will be submitted for publication in a peer reviewed journal.
Supporting Information: Study Protocol, ICF
Time Frame: Within one year
Access Criteria: Access to detailed information and IPD will be upon request. The PI and project team will evaluate the request based on the submission of an official request with details on what, why and how.

REFERENCES:
- [Derived] van Hoorn EGM, van Dijk PR, Prins JR, Lutgers HL, Hoogenberg K, Erwich JJHM, Kooy A. Pregnancy Outcomes: Effects of Metformin (POEM) study: a protocol for a long-term, multicentre, open-label, randomised controlled trial in gestational diabetes mellitus. BMJ Open. 2022 Mar 30;12(3):e056282. doi: 10.1136/bmjopen-2021-056282. PMID 35354633